CLINICAL TRIAL: NCT04488133
Title: A Phase 4 Study of Nusinersen (BIIB058) Among Patients With Spinal Muscular Atrophy Who Received Onasemnogene Abeparvovec
Brief Title: A Study to Learn About the Effect of Nusinersen (BIIB058) Given as Injections to Children With Spinal Muscular Atrophy (SMA) Who Were Previously Treated With Onasemnogene Abeparvovec (RESPOND)
Acronym: RESPOND
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 232SM404; 2020-003492-18 (EudraCT Number); 2023-505640-18 (Other: EU Trial Number)
Record Dates: First submitted 2020-07-20; First posted 2020-07-27 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Muscular Atrophy, Spinal
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — nusinersen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nusinersen 12 mg (Experimental): Participants will receive Nusinersen 12 milligrams (mg) via intrathecal (IT) injection as loading doses on Days 1, 15, 29, and 64 followed by maintenance doses, every 4 months, on Days 183, 302, 421, 540 and 659.
  Interventions: Drug: Nusinersen

INTERVENTIONS:
Drug: Nusinersen — Administered as specified in the treatment arm.
  Other Names: ISIS 396443; BIIB058; Spinraza

SUMMARY:
In this study, researchers will learn more about the use of nusinersen (BIIB058) in participants with spinal muscular atrophy (SMA). This study will focus on children under the age of 3 who were previously treated with the gene therapy onasemnogene abeparvovec but are still facing health challenges related to their disease.

The main goal of the study is to learn about the effect nusinersen has on muscle and movement ability (motor function). The main question researchers want to answer is:

- What score do participants have on the HINE Section 2 Motor Milestones test after treatment?

The Hammersmith Infant Neurological Examination (HINE) Section 2 Motor Milestones is an assessment that tests movements in different positions. This includes grasping, kicking, head control, rolling, sitting, crawling, standing, and walking.

Researchers will use a group of tests to study body movements, reflexes, balance, and coordination. They will also record if participants need help with breathing.

Researchers will also learn more about the safety of nusinersen. They will check participants for adverse events and changes in vital signs, heart tests, and laboratory tests including blood and urine tests.

The study will be done as follows:

* Participants will be screened to check if they can join the study.
* Each participant will receive 4 initial doses of 12 mg of nusinersen on Days 1, 15, 29, and 64 of the Treatment Period. Then, they will receive 12 mg doses once every 4 months.
* The total number of doses of nusinersen will be 9.
* Nusinersen will be given through a lumbar puncture, which involves injecting the drug into the fluid around the spinal cord in the lower back.
* The treatment period will last for up to 95 weeks (close to 2 years).
* There will be a follow-up safety period that lasts about 4 months.
* In total, participants will have up to 14 study visits. Participants will stay in the study for up to 115 weeks.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the clinical outcomes following treatment with nusinersen in participants with spinal muscular atrophy (SMA) who previously received onasemnogene abeparvovec.

The secondary objectives of this study are to evaluate the safety and tolerability; clinical outcomes and pharmacodynamics (PD) of nusinersen treatment in participants with SMA who previously received onasemnogene abeparvovec.

ELIGIBILITY:
Key Inclusion Criteria:

For all participants:

* Genetic documentation of 5q SMA homozygous gene survival motor neuron 1 (SMN1) deletion or mutation, or compound heterozygous mutation
* SMN2 copy number of ≥1
* ≤36 months of age at the time of first Nusinersen dose
* Must have previously received onasemnogene abeparvovec per the approved label or local/regional regulations ≥2 months prior to first Nusinersen dose
* Must have suboptimal clinical status per the Investigator

Additional Criteria for Subgroups A and B:

* <300 days of age at the time of first Nusinersen dose
* SMN2 copy number of 2

Additional Criteria for Subgroup A:

* SMA symptom onset ≤4 months (120 days) of age
* Must have received intravenous (IV) onasemnogene abeparvovec at >6 weeks to ≤6 months (43 days to 180 days) of age
* Must have received IV onasemnogene abeparvovec after SMA symptom onset

Additional Criteria for Subgroup B:

* Must have received IV onasemnogene abeparvovec at ≤6 weeks (42 days) of age

Key Exclusion Criteria:

For all participants:

* Prior exposure to Nusinersen
* Ongoing severe or serious AEs related to onasemnogene abeparvovec
* Treatment with an investigational drug, biological agent, or device within 30 days or 5 half-lives of the agent, whichever is longer, prior to study; any prior or current treatment with any survival motor neuron 2 (SMN2)-directed splicing modifier; prior antisense oligonucleotide treatment or cell transplantation; gene therapy for the treatment of SMA other than onasemnogene abeparvovec. Note: treatment with onasemnogene abeparvovec as part of an investigational study is allowed

Additional Criteria for Subgroups A and B:

* Weight-for-age is below the third percentile, based on WHO Child Growth Standards at the time of receiving onasemnogene abeparvovec. Adjustments for the gestational weight of premature babies enrolled in Subgroups A and B are allowed provided IV onasemnogene abeparvovec was dosed per the approved label or per local/regional regulations.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 2 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2025-10-09 (Actual); Study Completion 2025-10-09 (Actual)

PRIMARY OUTCOMES:
Total Hammersmith Infant Neurological Examination (HINE) Section 2 Motor Milestones Score | Up to Day 778
  Section 2 of the HINE is used to assess motor milestones of the participants. It is composed of 8 motor milestone categories: voluntary grasp (0 to 3), ability to kick in supine position (0 to 4), head control (0 to 2), rolling (0 to 3), sitting (0 to 4), crawling (0 to 4), standing (0 to 3), and walking (0 to 3). Total HINE score is the sum of points from each item and can range from 0 to 26, with higher scores depicting better level of ability.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to Day 778
  An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal assessment such as an abnormal laboratory value), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. An SAE is any untoward medical occurrence that at any dose results in death, in the view of the Investigator, places the participant at immediate risk of death, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, results in a birth defect or is a medically important event.
Number of Participants with Change from Baseline in Clinical Laboratory Parameters | Up to Day 778
Number of Participants with Change from Baseline in Electrocardiograms (ECGs) | Up to Day 778
Number of Participants with Change from Baseline in Vital Signs | Up to Day 778
Number of Participants who Achieved Motor Milestones as Assessed by World Health Organization (WHO) Criteria | Up to Day 778
  The motor milestones as defined by WHO criteria includes the following six test items: sitting without support, hands-and-knees crawling, standing with assistance, walking with assistance, standing alone, and walking alone.
Change from Baseline in Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders (CHOP INTEND) Score | Up to Day 778
  The CHOP INTEND test is designed to evaluate the motor skills of infants with significant motor weakness. It includes 16 items (capturing neck, trunk, and proximal and distal limb strength) structured to move from easiest to hardest with the grading including gravity eliminated (lower scores) to antigravity movements (higher scores). All item scores range from 0-4. The total score ranges from 0-64, with higher scores depicting better response.
Change from Baseline in Hammersmith Functional Motor Scale - Expanded (HFMSE) Score | Up to Day 778
  The HFMSE is a tool used to assess motor function in children with SMA. The original 20 item Hammersmith Functional Motor Scale (HFMS) was expanded to include 13 additional items to improve sensitivity for the higher functioning ambulant population. Participants will be asked to complete a specific movement and are then graded on the quality and execution of that movement. Higher scores indicate higher levels of motor ability. The overall score is the sum of the scores for all activities, with a maximum score of 66 with higher scores depicting better ability to perform activities.
Change from Baseline in Revised Upper Limb Module (RULM) Score | Up to Day 778
  The RULM is developed to assess upper limb functional abilities participants with SMA. This test consists of upper limb performance items that are reflective of activities of daily living. The RULM is scored from 0 to 37 points, with higher scores indicating better function.
Time to Death or Permanent Ventilation | Up to Day 778
  Permanent ventilation is defined as tracheostomy or ≥16 hours ventilation/day continuously for >21 days in the absence of an acute reversible event.
Change From Baseline in Cerebrospinal Fluid (CSF) Levels of Neurofilament Light Subunit (NF-L) | Up to Day 659
Change From Baseline in Plasma Levels of NF-L | Up to Day 778

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (15):
- United States (9):
  - Arkansas Children's Hospital Research Institute, Little Rock, Arkansas
  - Stanford Neuromuscular Research, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Oregon Health and Science University (OHSU), Portland, Oregon
  - Children's Hospital Philadelphia - Neurology, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
- Universitaetsklinikum Hamburg-Eppendorf, Hamburg, Germany
- Schneider Children's Medical Center, Petah Tikva, Israel
- Italy (2):
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, Milan
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
- Spain (2):
  - Hospital Sant Joan de Déu, Esplugues Del Llobregat, Barcelona
  - Hospital Universitario La paz, Madrid

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on http://clinicalresearch.biogen.com/
URL: https://vivli.org/

REFERENCES:
- [Derived] Proud CM, Finkel RS, Parsons JA, Masson R, Brandsema JF, Kuntz NL, Foster R, Li W, Littauer R, Sohn J, Fradette S, Youn B, Paradis AD; RESPOND Study Group. Open-label phase IV trial evaluating nusinersen after onasemnogene abeparvovec in children with spinal muscular atrophy. J Clin Invest. 2025 Sep 16;135(22):e193956. doi: 10.1172/JCI193956. eCollection 2025 Nov 17. PMID 40956616
- See also: SMA Europe — https://www.sma-europe.eu/
- See also: CureSMA — https://www.curesma.org/
- See also: Muscular Dystrophy Association — https://www.mda.org/disease/spinal-muscular-atrophy
- See also: Child Neurology Foundation — https://www.childneurologyfoundation.org/
- See also: Biogen Trial Link — https://www.biogentriallink.com/en-us/home.html